CLINICAL TRIAL: NCT00945607
Title: Guided Relaxation Training for the Reduction of Self-Reported Stress in Individuals With Newly Diagnosed Breast Cancer
Acronym: 09-IM-01
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trinitas Comprehensive Cancer Center (Other)
Collaborators: Aptium Oncology Research Network (Network)
Responsible Party: Carol Blecher, RN, MS, AOCN, APNC, Trinitas Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09-IM-01
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer
Keywords: Complementary Medicine; Alternative Medicine; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Relaxation Training (Experimental): Eligible subjects who have been randomized to the intervention arm will be scheduled for GRT introduction and training with a research staff member. The GRT sessions will consist of six weekly on-site sessions in which the subject is provided instructions and then allowed to listen to the GRT CD. Subjects will be instructed to conduct independent GRT sessions at home, twice daily, at least four hours apart, for the duration of the study. Subjects will also be instructed that on the days of one-on-one sessions with a research staff member at TCCC, that they will only be required to perform the independent session once at home.
  Subjects will be provided with a diary to record the date and time of each independent GRT session performed at home. Subjects will be instructed to bring their completed diary with them at each subsequent visit.
  Interventions: Other: GRT (Guided Relaxation Training)
- Standard of Care(SOC) (No Intervention): Eligible subjects who are randomized to the SOC arm will not receive the GRT sessions. During the six week treatment phase, these subjects will only receive SOC provided to all subjects newly diagnosed with breast cancer at TCCC. This consists of an education session with the nurse or nurse practitioner. In addition, they will also be provided with supportive care and symptom management as needed. This arm will also be provided with a diary to record their stress level at least twice daily.

INTERVENTIONS:
Other: GRT (Guided Relaxation Training) — Weekly on-site GRT sessions at the center in combination with twice daily independent GRT sessions at home.
  Arms: Guided Relaxation Training

SUMMARY:
The primary objectives of this study are to determine if the use of Guided Relaxation Training (GRT) during cancer treatment in individuals with newly diagnosed breast cancer increases their ability to cope as measured by the Coping Self-Efficacy Scale (CSES) and reduces their perceived stress as measured by the Perceived Stress Scale (PSS).

DETAILED DESCRIPTION:
This is a study of self-reported stress in individuals with newly diagnosed breast cancer. Subjects will be randomized to either the standard of care (SOC) arm or the intervention arm. The principle investigators will be blinded to the arm assignment. The intervention utilized will be six weekly on-site GRT sessions. In addition, subjects will be provided with a CD utilizing a standardized GRT script and music for home use twice daily during the study period. During the intervention period, they will also be provided with a diary and required to keep a record of date and time of CD utilization at home. The subjects will also be required to record their stress level before and after each of the two home sessions. The sessions must be at least 4 hours apart.

The SOC arm will consist of an education session with the nurse or nurse practitioner and supportive care / symptom management as needed. This group will also be required to keep a daily diary in which they record their stress levels twice daily, at intervals separated by at least 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand English
* At or between the ages of 18 and 75
* Newly diagnosed with breast cancer (within 12 weeks of study entry)
* Expected to receive chemotherapy and/or radiation
* Willingness to complete CSES, PSS-14 and FACIT-F scales
* Minimum score of 4 on the 0-10 Visual Analog Scale for stress
* Willingness to participate for the 18 week duration of study and follow-up
* Ability to travel to cancer center weekly specifically for on-site guided relaxation training sessions
* Access to a CD player

Exclusion Criteria:

* Cognitive or mental status affecting ability to follow directions
* Previous or current use of complementary therapies for their cancer diagnosis, except herbal supplements
* Brain metastasis
* Treatment for any other diagnosis of cancer within the previous 5 years
* Any condition that, in the opinion of the investigator might interfere with the subject's participation in the study, pose an added risk for the subject or confound the assessment of the subject

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Determining if the use of GRT during treatment in individuals newly diagnosed with breast cancer reduces their perceived stress. | Endpoint
Determining if the use of GRT during treatment in individuals newly diagnosed with breast cancer increases their coping ability. | Endpoint

SECONDARY OUTCOMES:
Determining the effects of GRT on vital signs and self-reported levels of fatigue. | End Point
Determining differences of perceived levels of stress among various racial and ethnic groups. | End Point

CONTACTS AND LOCATIONS:
Overall Officials: Carol S Blecher, RN, MS, AOCN, APNC, Principal Investigator — Trinitas Comprehensive Cancer Center; Sharon Kurtz, RN, BSN, C.Ht., Principal Investigator — Trinitas Comprehensive Cancer Center
Locations (1):
- Trinitas Comprehensive Cancer Center, Elizabeth, New Jersey, United States